CLINICAL TRIAL: NCT07099781
Title: Relation Between Shoulder Lateral Rotators Strength and Hand Grip Strength After Arthroscopic Bankart Repair Surgery
Brief Title: Relation Between Hand Grip and Shoulder Muscle Strength After Surgical Stabilization of Shoulder Dislocations
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdeltawab Mohamed Abdeltawab Hassoun, physiotherapist, Cairo University
Other Study IDs: PT.REC/012/005367
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Arthroscopic Bankart Repair; Arthroscopic Shoulder Surgery; Hand Grip Strength; Rotator Cuff Strength
Keywords: Shoulder Instability; Arthroscopic Bankart Repair; Lateral Rotator Strength; Hand Grip Strength

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: handheld dynamometer and hand grip dynamometer — using handheld dynamometer and hand grip dynamometer to test the strength of the hand grip and lateral rotators of the shoulder

SUMMARY:
To investigate the correlation between shoulder lateral rotators strength (LRS) and hand grip strength (HGS) at different shoulder positions in patients following arthroscopic Bankart repair surgery for anterior shoulder instability.

DETAILED DESCRIPTION:
Anterior shoulder instability is a common clinical problem with a high incidence rate in athletes (Zacchilli and Owens., 2010). It may be a result of anterior force trauma to elevated, horizontally abducted, and externally rotated shoulder. In this position, stability is provided by the subscapularis, GH ligaments (particularly the anterior band of the inferior ligament), and the long head of the biceps (Ladd et al., 2021b). A high energy trauma may affect these structures, along with the attachment of the anterior capsule and glenoid labrum (Bankart lesion) (Ladd et al., 2021a) Traditionally, patients with first-time dislocation are managed conservatively however, the recurrence rate is high especially in the teenagers and younger population (Polyzois et al. 2016). in case of recurrent dislocation, surgical repair of the affected structures is performed either by open or arthroscopic approach (Kane et al., 2015).

After surgery, dynamic stability of the shoulder is important to ensure the repaired capsule, anteroinferior labrum and/or the inferior glenohumeral ligament are not vigorously stressed and compromised during daily living activities (Mueller et al., 2005) The muscles responsible for shoulder rotation serve as active stabilizers for the glenohumeral joint, and regaining strength in these muscles is crucial for stabilizing the joint during the recovery process after surgery (Edouard et al., 2012). In a previous study, researchers examined the progression of rotational muscle strength before and after open Bankart and modified Bristow procedures. The findings indicate that adequate muscle strength can be achieved six months post-surgery. Furthermore, the strength of these rotational muscles is closely linked to shoulder function and could serve as a useful indicator of glenohumeral instability following surgery (Amako et al., 2008).10 A cohort study found that after 4-8 months of postoperative Bankart repair, about 74% of patients regained their baseline range of motion and strength (Buckwalter V et al., 2018).

In a 13-year follow-up study, it was found that patients with less than 6 months of postoperative rehabilitation after arthroscopic Bankart repair surgery had an increased rate of recurrent dislocation (Aboalata et al., 2017).

Many studies found a positive correlation between hand gripping activity and rotator cuff muscle activity in healthy subjects. It was found that hand loading induces an elevation in intramuscular pressure within the supraspinatus (SSP) and infraspinatus (ISP) muscles (L. V. Roberts et al., 2008; Shenouda and El-Tokhy., 2014).

Previous literature advocates a relation between grip strength and the overall strength of the upper body, as well as it serves as an objective indicator of upper extremity function (Vaishya et al., 2024). Other studies have shown a positive correlation between isometric hand grip strength and isokinetic peak torque and work of the shoulder stabilizing muscles (Mandalidis and O'Brien 2010; Nascimento et al., 2012). This relationship suggests that a stable proximal shoulder girdle is necessary to facilitate optimal recruitment of distal muscles and effective transmission of force along the myofascial pathways (Huijing and Baan., 2003).

There are different mechanisms through which handgrip exercises elevate shoulder muscle activity. It was observed that the rotator cuff muscles, particularly the SSP and ISP, are more impacted by hand loading due to their role as stabilizers of the shoulder joint compared to muscles responsible for elevation such as the deltoid (D. R. Lee and Kim., 2016). Given that, maintaining stability of the glenohumeral joint (GHJ) is a primary function of the SSP and ISP, it is logical to anticipate an increase in their activity during hand activities to uphold joint stability (Blache et al., 2017).

Previous literature found that hand grip strength can be quantified by measuring the amount of static force that the hand can apply on the hand grip dynamometer that provides an objective index of the functional integrity of the upper extremity (Massy-Westropp et al., 2011). Another study showed that grip strength can be reliably used to assess the function of the lateral rotators of the shoulder in normal individuals (Horsley et al., 2016).

Up to author best knowledge, there is limited literature considering the correlation between hand grip strength and shoulder lateral rotator strength in patients with post Bankart repair surgery. Therefore, this study aims to assess the relation between hand grip strength and shoulder lateral rotators strength in various shoulder positions in patients who have undergone arthroscopic Bankart repair surgery six months postoperatively

ELIGIBILITY:
Inclusion Criteria:

1. Patients with arthroscopic Bankart repair surgery.
2. Patients have passed 6 months after surgery.
3. Patients have not surpassed 12 months from surgery
4. Age of the patient ranged from 18 to 40 years to avoid including people with potential degenerative rotator cuff tears.
5. Patients immediately started physical therapy program after surgery for 6 months.
6. Nearly or complete full ROM.
7. Absence of shoulder pain.
8. Normal contralateral arm without previous surgeries.

Exclusion Criteria:

1. Other associated surgeries such as slap repair or large humeral bone defect requiring remplissage.
2. Moderate to severe shoulder pain.
3. Incomplete ROM.
4. Presence of nerve injury after the initial trauma.
5. Past history of other previous surgeries on the affected limb.
6. Any surgery or musculoskeletal disorder related to the neck or the contralateral upper limb.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 15 patients aged 18 to 40 years Who underwent arthroscopic Bankart repair surgery
  Recruited from the outpatient physical therapy unit at International Mansoura Hospital
  Assessed 6 to 12 months postoperatively
  All had undergone a standardized 6-month physical therapy program
  Inclusion criteria ensured full or nearly full ROM and absence of shoulder pain
  Patients had no other musculoskeletal or neurological impairments affecting the shoulder or contralateral upper limb.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Correlation between shoulder lateral rotator strength (LRS) and hand grip strength (HGS) | 6-12 months post arthroscopic bankart repair
  LRS and HGS will be measured isometrically using handheld dynamometer and hand grip dynamometer in three standardized shoulder positions. The correlation between these two variables will be analyzed to assess the neuromuscular relationship postoperatively.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of physical therapy, Cairo University, Cairo
  - Faculty of physical therapy, Cairo University, Giza

REFERENCES:
- [Result] Brophy RH, Marx RG. The treatment of traumatic anterior instability of the shoulder: nonoperative and surgical treatment. Arthroscopy. 2009 Mar;25(3):298-304. doi: 10.1016/j.arthro.2008.12.007. PMID 19245994
- [Result] Bottoni CR, Wilckens JH, DeBerardino TM, D'Alleyrand JC, Rooney RC, Harpstrite JK, Arciero RA. A prospective, randomized evaluation of arthroscopic stabilization versus nonoperative treatment in patients with acute, traumatic, first-time shoulder dislocations. Am J Sports Med. 2002 Jul-Aug;30(4):576-80. doi: 10.1177/03635465020300041801. PMID 12130413
- [Result] Bonazza NA, Liu G, Leslie DL, Dhawan A. Trends in Surgical Management of Shoulder Instability. Orthop J Sports Med. 2017 Jun 28;5(6):2325967117712476. doi: 10.1177/2325967117712476. eCollection 2017 Jun. PMID 28695137
- [Result] Blackburn TA, Guido JA. Rehabilitation after ligamentous and labral surgery of the shoulder: guiding concepts. J Athl Train. 2000 Jul;35(3):373-81. PMID 16558650
- [Result] Su CY, Lin JH, Chien TH, Cheng KF, Sung YT. Grip strength in different positions of elbow and shoulder. Arch Phys Med Rehabil. 1994 Jul;75(7):812-5. PMID 8024431
- [Result] Steenbrink F, de Groot JH, Veeger HE, Meskers CG, van de Sande MA, Rozing PM. Pathological muscle activation patterns in patients with massive rotator cuff tears, with and without subacromial anaesthetics. Man Ther. 2006 Aug;11(3):231-7. doi: 10.1016/j.math.2006.07.004. PMID 16890886
- [Result] Boileau P, Villalba M, Hery JY, Balg F, Ahrens P, Neyton L. Risk factors for recurrence of shoulder instability after arthroscopic Bankart repair. J Bone Joint Surg Am. 2006 Aug;88(8):1755-63. doi: 10.2106/JBJS.E.00817. PMID 16882898
- [Result] Blache Y, Begon M, Michaud B, Desmoulins L, Allard P, Dal Maso F. Muscle function in glenohumeral joint stability during lifting task. PLoS One. 2017 Dec 15;12(12):e0189406. doi: 10.1371/journal.pone.0189406. eCollection 2017. PMID 29244838
- [Result] Arner JW, Peebles LA, Bradley JP, Provencher MT. Anterior Shoulder Instability Management: Indications, Techniques, and Outcomes. Arthroscopy. 2020 Nov;36(11):2791-2793. doi: 10.1016/j.arthro.2020.09.024. PMID 33172578
- [Result] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Result] Amako M, Imai T, Okamura K. Recovery of shoulder rotational muscle strength after a combined Bankart and modified Bristow procedure. J Shoulder Elbow Surg. 2008 Sep-Oct;17(5):738-43. doi: 10.1016/j.jse.2008.01.145. Epub 2008 Jun 16. PMID 18558501
- [Result] Amako M, Arino H, Tsuda Y, Tsuchihara T, Nemoto K. Recovery of Shoulder Rotational Muscle Strength After Arthroscopic Bankart Repair. Orthop J Sports Med. 2017 Sep 27;5(9):2325967117728684. doi: 10.1177/2325967117728684. eCollection 2017 Sep. PMID 28989939
- [Result] Alizadehkhaiyat O, Fisher AC, Kemp GJ, Vishwanathan K, Frostick SP. Shoulder muscle activation and fatigue during a controlled forceful hand grip task. J Electromyogr Kinesiol. 2011 Jun;21(3):478-82. doi: 10.1016/j.jelekin.2011.03.002. Epub 2011 Apr 2. PMID 21459609
- [Result] Alexander CM, Miley R, Harrison PJ. Functional modulation of shoulder girdle stability. Exp Brain Res. 2005 Mar;161(4):417-22. doi: 10.1007/s00221-004-2083-y. Epub 2004 Oct 21. PMID 15502981
- [Result] AlAnazi A, Alghadir AH, Gabr SA. Handgrip Strength Exercises Modulate Shoulder Pain, Function, and Strength of Rotator Cuff Muscles of Patients with Primary Subacromial Impingement Syndrome. Biomed Res Int. 2022 Aug 30;2022:9151831. doi: 10.1155/2022/9151831. eCollection 2022. PMID 36082154
- [Result] Aboalata M, Plath JE, Seppel G, Juretzko J, Vogt S, Imhoff AB. Results of Arthroscopic Bankart Repair for Anterior-Inferior Shoulder Instability at 13-Year Follow-up. Am J Sports Med. 2017 Mar;45(4):782-787. doi: 10.1177/0363546516675145. Epub 2016 Nov 24. PMID 27872125